CLINICAL TRIAL: NCT05534178
Title: Machine Learning Model to Predict Hospital Length of Stay (HOLS) and Mortality After Discharge in Hospitalized Oncologic Patients [Plantology Database]: a Multicenter Cross-validation Study
Brief Title: Machine Learning Model to Predict HOLS and Mortality After Discharge in Hospitalized Oncologic Patients
Acronym: PLANTOLOGY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital del Mar (Other)
Responsible Party: Principal Investigator, Oriol Mirallas, Principal Investigator, Vall d'Hebron Institute of Oncology
Other Study IDs: VHIO1601
Record Dates: First submitted 2022-03-27; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Solid Tumor; Nutrition Related Neoplasm/Cancer; Comorbidities and Coexisting Conditions; Mental Status Change; Artificial Intelligence; Oncology; Tumor; Quality of Life
Keywords: Hospitalization; Oncologic patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to understand which are the most relevant parameters at admission which may allow to predict the hospital length of stay (HOLS) and mortality after discharge of oncologic hospitalized patients.

This is the first multicentric prospective observational study that tries to understand the complexity of the hospitalized oncologic patients. A comprehensive analysis will be performed with the help of the nutrition, nursery, internal medicine and oncology teams.

DETAILED DESCRIPTION:
BACKGROUND:

Cancer is the second leading cause of death worldwide and is responsible for about 18.1 million new cases and 9.6 million deaths in 2018 alone according to the International Agency for Research on Cancer. Cancer is anticipated to rank as the leading cause of death and the most important barrier to increasing life expectancy in every country of the world in the mid-21st century1. The economic impact of cancer is significant. The annual economic cost of cancer in 2010 was estimated at approximately US$ 1.16 trillion. The reasons are complex but both cancer incidence and mortality are increasing worldwide due to aging and increasing risk factors for cancer, several of which are associated with socioeconomic development. Cancer will probably soon reach the top leading cause of death due to the rapid population growth and the declines in mortality rates by stroke or coronary heart disease in many developed countries.

Cancer patients often require inpatient care due to treatment toxicities, complications from cancer such as thrombosis, illness not related to the disease itself or terminally ill patients. Among these individuals, their treatment should balance prolongation of survival and maximization of the quality of remaining life. However, hospitalization is a stressful event for individuals with advanced cancer and their caregivers. Hospitalization often antagonizes these goals, contributing to the high cost of cancer care, worsens survival, and is increasingly recognized as poor-quality cancer care. Thus, interventions that reduce unnecessary hospitalizations, or shorten them, will likely improve quality of life and reduce costs.

Some studies relate malnutrition, which presents a marked sarcopenia and loss of lean mass, with prolonged hospitalization, reduced response to treatment, a worse overall survival and impaired quality of life. A study published in 2007 found that lung cancer patients had a longer hospitalization and required inpatient hospital treatment more frequently than any other type of tumor. Moreover, in the surgical setting there have been studies linking preoperative opioid usage and increased opioid doses with increased length of stay. Based on this data, there have been protocols developed like the ERAS (Enhanced recovery after surgery) applied first to colorectal cancer and now being tested in other settings like head and neck and gynecologic tumors, showing that it is possible to reduce opioid use with good pain control and a statistically significant shorter average length of stay.

Prognostic factors for oncologic patients after surgery or curative systemic treatment have been described, but there is no solid evidence on which combination of parameters predict mortality after hospitalization of metastatic cancer patients under active treatment. A potential solution to improve this scenario might be nutritional support to malnourished cancer patients that also has proven to be effective in shorten hospital stay and improve survival, or community based palliative care interventions that are proven to improve quality of life and reduce costs of terminally ill patients. Thus, a prognostic tool would be useful to help physicians adjust medical interventions for hospitalized cancer patients.

To the best of our knowledge, this is the first study that examines independent clinical, psychological, nutritional status, and laboratory characteristics of oncologic patients in order to grasp a comprehensive picture of what factors play a role in the length of stay, mortality, and quality of life.

MEANING The investigators pretend with this work to fill a gap of knowledge in the oncology field through a prospective study. The investigators would like to measure the effect of hospitalization on oncologic patients after discharge and how clinical and laboratory parameters at admission may be able to predict HOLS and 30-day mortality after discharge. The investigators would also like to validate the different scales already published to assess nutritional status, psychological status, quality of life or prediction of rehospitalization for oncologic patients in all-in-one study.

This study will hopefully be able to develop a predictive tool at admission to help physicians adjust medical interventions and detect possible actions that will need to be implemented during hospitalization in order to improve the overall survival and quality of life of our patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years-old.
* Histological cancer confirmation.
* Hospitalization in oncology ward.

Exclusion Criteria:

* <18 years-old.
* Not histological malignancy confirmed.
* Less than 24 hours in the hospital.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All oncologic patients that require hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Predict Mortality | 30 days after discharge
  Mortality at 30-day after discharge
Predict hospital length of stay | Through study completion, an average of 3 years
  Number of days hospitalized

SECONDARY OUTCOMES:
Measure the impact of Anxiety and Depression | Within 24 hours of admission
  Hospital Anxiety and Depression Scale (HADS). Minimum: 0 Maximum: 21. More than 12 points is clinical significant for depression or anxiety [0-7 = Normal; 8-10 = Borderline; abnormal (borderline case)] 11-21 = Abnormal (case)
Measure the impact of Quality of life (QoL) | Within 24 hours of admission
  EORTC QLQ-C30 Minimum: 30 Maximum: 126. More punctuation, worse QoL
Validate standardized test HOSPITAL score: Risk of readmission | Evaluated at discharge through study completion, an average of 3 years. The outcome is the probability of readmission within the first 30 days after discharge.
  HOSPITAL Score; higher score, more risk of readmission. Min: 0 points. Max: 13 points. Measures: Risk of potentially avoidable 30-day readmission.
Sarcopenia Assessment | Within 24 hours of admission and 24 hours before discharge through study completion, an average of 3 years
  Chair test is performed by the number of stands a person can complete in 30 seconds. Results depend on sex and age, the more the better and screens for sarcopenia.
Sarcopenia Test | Within 24 hours of admission and 24 hours before discharge through study completion, an average of 3 years
  Hand grip test; the more power the better using a hand-held dynamometer. It screens for sarcopenia. A poor performance is 20 to 22kg of power, a below average performance is 23 to 35kg of power, an average performance is 26 to 29kg of power, and an above average performance is 30 to 33kg of power.
Nutrition Assessment | Within 24 hours of admission and 24 hours before discharge through study completion, an average of 3 years
  Intake compliance of food served (100%, 75%, 50%, 25% and 0% of the food served in each meal.
Opioids Intake | Within 24 hours of admission and 24 hours before discharge through study completion, an average of 3 years
  Quantity of morphine equivalent in mg per day at admission and at discharge
Tumor Characteristics and Comorbidities | Within 24 hours of admission through study completion, an average of 3 years
  Tumor type, oncologic treatment during the last 6 months, comorbidities measured through the Charlson score (Age, <50years 0 points, 50-59years 1 point, 60-69 years 2 points, 70-79 years 3 points, =>80 years, 4 points, Prior myocardial infarction 1 point; congestive heart failure 1 point; peripheral vascular disease 1point; Cerebrovascular disease 1 point; Dementia 1 point; Chronic pulmonary disease 1 point; Rheumatologic disease 1 point; Peptic ulcer disease 1 point; Mild liver disease 1 point; Diabetes 1 point; Cerebrovascular (hemiplegia)event 2 points; Moderate-to-severe renal disease 2 points; Cancer without metastases 2 points; Leukemia 2 points; Lymphoma 2 points; Moderate to severe liver disease 3 points; Metastatic Solid tumor 6 points; Acquired immune deficiency syndrome (AIDS; 6 points). Max 37 points. Min 0 points. The higher the score, the more comorbidities and worse survival.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Mirallas, MD, Principal Investigator — Vall d'Hebron University Hospital
Locations (3):
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with all the participants of the study
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year
Access Criteria: Principal investigators and sub-investigators

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Brooks GA, Cronin AM, Uno H, Schrag D, Keating NL, Mack JW. Intensity of Medical Interventions between Diagnosis and Death in Patients with Advanced Lung and Colorectal Cancer: A CanCORS Analysis. J Palliat Med. 2016 Jan;19(1):42-50. doi: 10.1089/jpm.2015.0190. Epub 2015 Nov 24. PMID 26600474
- [Result] Manzano JG, Luo R, Elting LS, George M, Suarez-Almazor ME. Patterns and predictors of unplanned hospitalization in a population-based cohort of elderly patients with GI cancer. J Clin Oncol. 2014 Nov 1;32(31):3527-33. doi: 10.1200/JCO.2014.55.3131. Epub 2014 Oct 6. PMID 25287830
- [Result] Earle CC, Park ER, Lai B, Weeks JC, Ayanian JZ, Block S. Identifying potential indicators of the quality of end-of-life cancer care from administrative data. J Clin Oncol. 2003 Mar 15;21(6):1133-8. doi: 10.1200/JCO.2003.03.059. PMID 12637481
- [Result] Whitney RL, Bell JF, Tancredi DJ, Romano PS, Bold RJ, Joseph JG. Hospitalization Rates and Predictors of Rehospitalization Among Individuals With Advanced Cancer in the Year After Diagnosis. J Clin Oncol. 2017 Nov 1;35(31):3610-3617. doi: 10.1200/JCO.2017.72.4963. Epub 2017 Aug 29. PMID 28850290

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT05534178/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT05534178/ICF_001.pdf